CLINICAL TRIAL: NCT05179746
Title: Adjunctive Benefit of Electrolytic Cleaning on Non-surgical Treatment of Peri-implantitis. A 1-year Randomized Controlled Clinical Trial.
Brief Title: Adjunctive Benefit of Electrolytic Cleaning on Non-surgical Treatment of Peri-implantitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Vanessa Rocha Rodrigues, Dr, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Electrolytic cleaning
Record Dates: First submitted 2021-12-03; First posted 2022-01-05 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Peri-Implantitis
Keywords: treatment of peri-implantitis; electrolytic cleaning
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With electrolytic cleaning (Active Comparator): Mechanical debridement with ultrasonics (plastic tip) and plastic curettes
  Interventions: Device: Implants are decontaminated with electrolytic cleaning
- Without electrolytic cleaning (Placebo Comparator): Mechanical debridement with ultrasonics (plastic tip) and plastic curettes
  Interventions: Device: Implants are decontaminated without electrolytic cleaning

INTERVENTIONS:
Device: Implants are decontaminated with electrolytic cleaning — Implants are decontaminated with electrolytic cleaning
  Arms: With electrolytic cleaning
Device: Implants are decontaminated without electrolytic cleaning — Implants are decontaminated without electrolytic cleaning
  Arms: Without electrolytic cleaning

SUMMARY:
Evaluate the outcomes of non-surgical therapy of peri-implantitis with the adjunctive use of electrolytic cleaning (Galvo Surge®).

The proposed protocol, focused on the non-surgical treatment of peri-implantitis, will result in a higher percentage of subjects with disease resolution (probing depts ≤ 5mm, absence of BOP and/or SOP and no further bone loss) at 1 year of follow-up.

DETAILED DESCRIPTION:
The adjunctive use of electrolytic cleaning (Galvo Surge®) in the non-surgical treatment of peri-implantitis will result in a higher reduction of probing depth than the control group.

The adjunctive use of electrolytic cleaning (Galvo Surge®) in the non-surgical treatment of peri-implantitis will result in a higher radiographic bone fill of the peri-implant defect than the control group.

The adjunctive use of electrolytic cleaning (Galvo Surge®) in the non-surgical treatment of peri-implantitis will result in a lower count of peri-implant pathogens than the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Partially edentulous patients, rehabilitated with at least one dental implant in the maxilla or mandible;
2. Presence of Peri-implantitis;
3. No implant mobility;
4. Treated periodontal disease;
5. No systemic diseases that could influence the outcome of the therapy (i.e. uncontrolled diabetes, osteoporosis, bisphosphonate medication).
6. Non-smoker or light smoking status in smokers (<10 cigarettes/day).

Exclusion Criteria:

(1) Pregnant, lactating women and non-collaborating patients will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | Assessing the change of probing pocket depth from baseline at 3 months, 6 months and 12 months
  Will be calculated as the distance from the gingival peri-implant margin to the bottom of the peri-implant pocket (Mombelli & Lang, 1994).
Recession | Assessing the change of recession from baseline at 3 months, 6 months and 12 months
  will be measured as the distance from the free marginal mucosa to the most apical portion of the crown.
Clinical attachment level | Assessing the change from clinical attachment level from baseline at 3 months, 6 months and 12 months
  will be calculated as the sum of PPD and REC (distance from the most apical portion of the crown to the bottom of the periodontal pocket)
Bleeding on probing | Assessing the change from bleeding on probing from baseline at 3 months, 6 months and 12 months
  will be assessed dichotomously in six sites per implant (Heitz-Mayfield, 2008).
Radiographic Parameters | Assessing the change of the radiographic parameters from baseline at 3 months, 6 months
  Radiographic analysis through orthopantomography, periapical intraoral radiographs according to the parallelometric technique (using a silicone bite record so that the radiographs are parallelized and comparable to each other in different timepoints, checking in millimeters the increase or decrease in bone loss).

SECONDARY OUTCOMES:
Microbiological Parameters | Assessing the change of the microbiological parameters from baseline at 3 months, 6 months
  A sterilized paper tip from the microbiological kit will be introduced in the periimplantitis pocket, remaining in the same position for 10 seconds. After collecting the sample, the paper tip will be placed in an individual transfer tube, properly identified. Afterwards, the sample will be sent to the laboratory, where a polymerase chain reaction (PCR) test is performed to identify the following bacteria - A. actinomycetemcomitans, T. forsythia, T. denticola, P. gingivalis, P. intermedia and F. nucleatum.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Ribeiro-Amaral, Dr, Principal Investigator — University of Lisbon; Paulo Macaranhas, PhD, Study Director — University of Lisbon; Vanessa Rocha Rodrigues, Dr, Study Chair — University of Lisbon; Susana Noronha, PhD, Study Director — University of Lisbon

IPD SHARING:
Plan to Share IPD: No